CLINICAL TRIAL: NCT01681849
Title: Neural Circuits in Women With Abuse and Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, J. Douglas Bremner, M.D., Professor of Psychiatry and Radiology, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00000857; R01MH056120 (NIH)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: PTSD
Keywords: PTSD; childhood abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paroxetine Group (Experimental): Women who have experienced early childhood abuse and have PTSD will be randomized in a double blind fashion to receive paroxetine for a three month period followed by an open label phase of three months.
  Interventions: Drug: Paroxetine; Other: Positron Emission Tomography (PET) Imaging
- Placebo Group (Placebo Comparator): Women who have experienced early childhood abuse and have PTSD will be randomized in a double blind fashion to receive placebo for a three month period followed by an open label phase of paroxetine for three months.
  Interventions: Drug: Placebo; Drug: Paroxetine; Other: Positron Emission Tomography (PET) Imaging
- PTSD Negative (Other): Women who have experienced early childhood abuse and do not have PTSD will serve as a control group and complete baseline assessments. They do not undergo intervention therefore they are assessed at baseline only.
  Interventions: Other: Positron Emission Tomography (PET) Imaging

INTERVENTIONS:
Drug: Placebo — Following a three month double blind phase, subjects will be treated with open label paroxetine at a variable dosage of 10-40 mg to reach individual therapeutic levels for three months.
  Arms: Placebo Group
Drug: Paroxetine — Following a three month double blind phase, subjects will be treated with open label paroxetine at a variable dosage of 10-40 mg to reach individual therapeutic levels for three months.
  Other Names: Paxil
  Arms: Paroxetine Group; Placebo Group
Other: Positron Emission Tomography (PET) Imaging — Participants will undergo positron emission tomography (PET) imaging of the brain with O-15 radiolabelled water with exposure to traumatic scripts

SUMMARY:
The purpose of this study was to assess the effects of the medication paroxetine on symptoms of posttraumatic stress disorder (PTSD) and the brain in women with a history of PTSD related to childhood abuse. The hypothesis is that paroxetine will result in an improvement in PTSD symptoms accompanied by changes in brain functional response to reminders of childhood trauma.

DETAILED DESCRIPTION:
The main purpose of this study was to look at the effects of paroxetine on PTSD symptoms and brain function in women with posttraumatic stress disorder (PTSD) related to childhood abuse. Participants underwent baseline assessment with of PTSD symptoms measured with the Clinician Administered PTSD Scale (CAPS) and brain function during exposure to traumatic scripts of childhood abuse. Participants then were treated in a randomized double-blind fashion with paroxetine or placebo for three months, followed by a repeat of these assessments.

Specific Aims of this proposal were therefore to:

* Assess the effects of paroxetine on PTSD symptoms
* Assess the effects of paroxetine on brain function in conjunction with exposure to traumatic scripts using positron emission tomography (PET) with O-15 water

ELIGIBILITY:
Inclusion Criteria:

* Subjects meet criteria for current PTSD as determined by the Structured Clinical Interview for DSMIV (SCID) interview for PTSD and the Clinician Administered PTSD Scale (CAPS) and have a score of greater than 60 on the CAPS
* history of penetrative sexual abuse which occurred once a month or more, for a period of greater than a year at some time between the ages of 4-13, as assessed by the Early Trauma Inventory (ETI)
* are free of psychotropic medication for four weeks before the study (subjects will not be taken off of medication for the purpose of the study).
* Non-PTSD subjects will be included based on the same criteria with the exception that they do not meet criteria for PTSD.

Exclusion Criteria:

* a history of shrapnel or other foreign bodies which would preclude MRI scanning
* meningitis
* traumatic brain injury
* neurological disorder or organic mental disorder
* history of loss of consciousness
* alcohol abuse or substance abuse or dependence based on the SCID within the past 24 months
* positive pregnancy test as measured by a serum beta-HCG or urine pregnancy test on the morning of the PET scan. Women will be counseled about the risks of pregnancy during the course of the study
* current or lifetime history of schizophrenia, schizoaffective disorder, or bulimia, based on the SCID
* a history of serious medical or neurological illness, such as cardiovascular, gastrointestinal, hepatic, renal, neurologic or other systemic illness
* evidence of a major medical or neurological illness on physical examination or as a result of laboratory studies (CBC, BUN, creatinine, blood sugar, electrolytes, liver and thyroid function tests, urinalysis, and EKG)
* positive urine toxicology screen
* history of ongoing violence such as domestic abuse as measured by the ETI-lifetime
* post-menopausal status as measured by menstrual history.
* Non-PTSD subjects will additionally be excluded with current major depression or other major psychiatric disorder based on the SCID.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Bremner, MD, Principal Investigator — Professor
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Clinic and Emory University Hospitals from September 2006 to November 2013.
Pre-assignment Details: Of the 91 participants who were consented, 7 were excluded due to not meeting screening criteria.
Groups:
- Paroxetine Group: Women who have experienced early childhood abuse and have PTSD were randomized in a double blind fashion to receive paroxetine for a three month period followed by an open label phase of three months.
  Paroxetine: Following a three month double blind phase, subjects were treated with open label paroxetine at a variable dosage of 10-40 mg to reach individual therapeutic levels for three months.
  Positron Emission Tomography (PET) Imaging: Participants underwent positron emission tomography (PET) imaging of the brain with O-15 radiolabelled water while completing memory tasks.
- Placebo Group: Women who have experienced early childhood abuse and have PTSD were randomized in a double blind fashion to receive placebo for a three month period followed by an open label phase of paroxetine for three months.
  Placebo: Following a three month double blind phase, subjects were treated with open label paroxetine at a variable dosage of 10-40 mg to reach individual therapeutic levels for three months.
  Paroxetine: Following a three month double blind phase, subjects were treated with open label paroxetine at a variable dosage of 10-40 mg to reach individual therapeutic levels for three months.
  Positron Emission Tomography (PET) Imaging: Participants underwent positron emission tomography (PET) imaging of the brain with O-15 radiolabelled water while completing memory tasks.
- PTSD Negative: Women who have experienced early childhood abuse and do not have PTSD served as a control group and completed baseline assessments
  Positron Emission Tomography (PET) Imaging: Participants underwent positron emission tomography (PET) imaging of the brain with O-15 radiolabelled water while completing memory tasks.
Period: Overall Study
Arm/Group | Paroxetine Group | Placebo Group | PTSD Negative
Started | 15 | 13 | 56
Completed | 7 | 6 | 17
Not Completed | 8 | 7 | 39
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 33
Not completed — Lost to Follow-up | 3 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine Group | Placebo Group | PTSD Negative | Total
Number analyzed (Participants) | 15 | 13 | 56 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 56 | 84
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 56 | 84
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 56 | 84

OUTCOME MEASURES:

1. Primary Outcome: Mean Clinical Administered PTSD Scale for DSM-IV (CAPS) Score
Description: The CAPS is a 30-item questionnaire of PTSD symptomatology that provides continuous measures of symptom severity and frequency. CAPS-IV total symptom severity score is calculated by summing severity scores for the 17 DSM-IV PTSD symptoms. Each symptom is rated for severity based on frequency and intensity on a scale of 0-4 for a total possible severity score per symptom of 8. Criterion E (items 18-19) is duration of symptoms (minimum of one month to make the diagnosis). Items 20-30 are optional. CAPS score is based on items 1-17, CAPS score has a potential range of 0-136, with higher scores indicating greater severity of PTSD symptoms. CAPS was performed before and after treatment with paroxetine or placebo in PTSD patients.
Time Frame: Baseline, End of Study (Up to 52 Weeks)
Population: Data for participants who completed all study visits were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine Group | Placebo Group
Number analyzed (Participants) | 7 | 6
units on a scale
  Baseline | 31 (10) | 30 (5)
  End of Study (Up to 52 Weeks) | 20 (10) | 25 (6)

2. Secondary Outcome: Change in Brain Blood Flow Assessed by Statistical Parametric Mapping (SPM)
Description: Participants were exposed to traumatic scripts versus neutral scripts before and after treatment with paroxetine or placebo. Brain blood flow was measured using statistical parametric mapping (SPM) which analyzes brain imaging data sequences. Statistical Parametric Mapping software is only capable of producing a single z-score for each Arm/Group. Data for each participant can not be generated using this software and therefore are not available to summarize in the data table below. Regional blood flow was compared for stress and neutral conditions and before and after treatment with paroxetine or placebo. Higher z-scores indicate an increase in regional blood flow to the medial prefrontal cortex under stress conditions for the 3 month time point relative to baseline. Statistical Parametric Mapping software is only capable of producing a single z-score for each Arm/Group.
Time Frame: Baseline, 3 Months Post Treatment
Population: Statistical analyses yielded image data sets in which the values assigned to individual voxels correspond to the t-statistic of the difference in brain blood flow between conditions. Statistical images were displayed with values of z score units.
Measure: Number; unit: z-scores
Arm/Group | Paroxetine Group | Placebo Group
Number analyzed (Participants) | 7 | 6
z-scores | 22 | 2.68

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study and open label period (2 years). Adverse events were collected for all participants who began the study.
Groups:
- Paroxetine Group: Women who have experienced early childhood abuse and have PTSD will be randomized in a double blind fashion to receive paroxetine for a three month period followed by an open label phase of three months.
  Paroxetine: Following a three month double blind phase, subjects will be treated with open label paroxetine at a variable dosage of 10-40 mg to reach individual therapeutic levels for three months.
  Positron Emission Tomography (PET) Imaging: Participants will undergo positron emission tomography (PET) imaging of the brain with O-15 radiolabelled water while completing memory tasks.
- Placebo Group: Women who have experienced early childhood abuse and have PTSD will be randomized in a double blind fashion to receive placebo for a three month period followed by an open label phase of paroxetine for three months.
  Placebo: Following a three month double blind phase, subjects will be treated with open label paroxetine at a variable dosage of 10-40 mg to reach individual therapeutic levels for three months.
  Paroxetine: Following a three month double blind phase, subjects will be treated with open label paroxetine at a variable dosage of 10-40 mg to reach individual therapeutic levels for three months.
  Positron Emission Tomography (PET) Imaging: Participants will undergo positron emission tomography (PET) imaging of the brain with O-15 radiolabelled water while completing memory tasks.
- PTSD Negative: Women who have experienced early childhood abuse and do not have PTSD will serve as a control group and complete baseline assessments
  Positron Emission Tomography (PET) Imaging: Participants will undergo positron emission tomography (PET) imaging of the brain with O-15 radiolabelled water while completing memory tasks.
Arm/Group | Paroxetine Group | Placebo Group | PTSD Negative
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/56
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes